CLINICAL TRIAL: NCT02657798
Title: Resist: What Are the Mechanisms Involved in Depression and Antidepressant Resistance That Increase Cardiovascular Risk?
Brief Title: RESIST: Understanding the Role of Depression in Heart Disease
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0860
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva, peripheral blood mononuclear cells, blood serum, blood plasma, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Depressed patients taking sertraline: Patients with depression who have been randomised to the sertraline arm in the PANDA trial
- Depressed patients taking placebo: Patients with depression who have been randomised to the placebo arm in the PANDA trial
- Healthy controls: Healthy participants with no history of depression

SUMMARY:
This study will investigate the biological pathways involved in anti-depressant resistance that increase risk of cardiovascular disease in people with depression.

DETAILED DESCRIPTION:
Rationale: Depression is known to be associated with the development of cardiovascular disease and poorer prognosis after cardiac events, however the mechanisms that mediate these links are poorly understood. Inflammatory and neuroendocrine processes are thought to play an important role in this relationship. In addition, antidepressants have been shown to improve cardiac outcomes and have anti-inflammatory effects, whilst inflammation has been shown to be elevated in patients who do not respond to treatment. Several possible biomarkers for antidepressant resistance have also been demonstrated to be cardiovascular risk markers. These include acute phase inflammatory markers, such as interleukin-6 (IL-6), and hypothalamic-pituitary-adrenal axis (HPA) dysregulation.

Design: This will be conducted alongside a larger pharmacological trial, PANDA, where participants will be recruited from primary care and randomized to sertraline (SSRI) or placebo. The RESIST study will compare inflammatory cardiovascular risk factors between depressed patients taking sertraline, depressed patients taking placebo and healthy controls. This will be achieved by investigating the pharmacological effect of antidepressants on gene expression, glucocorticoid and mineralocorticoid receptor function and regulatory T cell (Treg) profiles.

ELIGIBILITY:
Inclusion Criteria:

* Depressed patients:

  * Meet ICD10 criteria from the Clinical Interview Schedule-Revised (CIS-R)

Exclusion Criteria:

* Depressed patients:

  * Are taking any anti-inflammatory drugs or drugs which interfere with HPA-axis function, endothelial function, circadian rhythm or any other pathways under investigation
  * Unable to read, understand and/or complete questionnaires
  * Other psychiatric disorders: psychosis, schizophrenia, bipolar disorder, mania, hypomania, dementia, and eating disorder
  * Vulnerable adults
* Healthy controls:

  * Have a history of depression
  * Are taking any anti-inflammatory drugs or drugs which interfere with HPA-axis function, endothelial function or circadian rhythm or any other pathways under investigation
  * Unable to read, understand and/or complete questionnaires
  * Other psychiatric disorders: psychosis, schizophrenia, bipolar disorder, mania, hypomania, dementia, and eating disorder
  * Vulnerable adults

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Depressed patients will be recruited from the PANDA trial. Healthy controls will be recruited from primary care.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Candidate gene expression | 6 weeks
  Levels of RNA expression for genes associated with cardiovascular risk
Glucocorticoid and mineralocorticoid receptor function | 6 weeks
  Glucocorticoid and mineralocorticoid inhibition of lipopolysaccharide (LPS)-stimulated IL-6 levels.
Regulatory T-cell profiles | 6 weeks
  Measurement of percentages of leukocyte subsets

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Lewis, Principal Investigator — UCL
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No